CLINICAL TRIAL: NCT01287468
Title: Academia Sinica Investigator Award 2010
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ning-Sun Yang, Agricultural Biotechnology Research Center, Academia Sinica
Other Study IDs: 99052
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: phytomedicines; breast cancer; stromal fibroblasts; MDSCs; functional mechanism
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
Over the past five years, a spectrum of studies has shown that the stromal cell populations surrounding or embedding cancer cells in a variety of different tumor types are intrinsically involved in the mechanisms affecting tumor growth and metastasis. Among these cells, fibroblasts and myeloid derived suppressor cells (MDSCs) have been shown to play key roles in the regulation of tumor cell behaviors, via differential gene expression, regulation and secretion of specific chemokines (e.g., RANTES, CXCL12 and CXCL14), cytokines (e.g., TNF-α, IL-1β, NF-κB) and control by inflammatory and immunomodulatory cells, molecules or potent growth factors. Of particular interest is that the various stromal immune cells (dendritic cells and T cells) and inflammatory MDSCs found in primary and metastatic tumors behave very differently from those present in normal or non-cancerous counterpart tissues. In light of these "new understandings" in cancer biology, the investigators believe that systematic and innovative approaches to further research are very much needed in Taiwan and at our Academy. Here the investigators propose to investigate the tumor suppressive effect of anti-inflammatory phytomedicines on regulation of stromal immune cells and fibroblasts in breast cancers. The investigators will employ the TS/A and 4T1 mouse mammary carcinoma system to conduct an in vivo study of several specific candidate phytomedicines (cytopiloyne, Wedelia chinensis, shikonin, emodin and others that the investigators have already identified as conferring anti-inflammation related activities) for inhibition of TS/A and 4T1 tumor growth and specific effects on inflammation-associated, cellular and molecular functions of stromal immune cells, fibroblasts and MDSCs. When potent and specific anti-tumor effects are detected, the investigators will extend our study to a three-dimensional collagen/Matrigel culture system for ex-vivo study focusing on the stromal cell-mediated or -associated anti-tumor effects of TS/A or 4T1 cells, using the "organoid" tissue culture systems the investigators have previously developed in our laboratory (JNCI, 1979; Cancer Res., 1981). The investigators will establish reconstituted TS/A or 4T1 tumor cells with the stromal immune cells in a co-cultivation system. When the investigators have achieved demonstrable success, the investigators will extend the mouse system to human breast cancers (including primary and metastatic tumors) by a close collaboration (which the investigators have already established) with Drs.

DETAILED DESCRIPTION:
Ji-Hong Jhu (朱紀洪, Hospital President, M.D./surgeon) and Huey-Kong Sytwu (司徒惠康, M.D., Ph.D.) at the National Defense University Hospital. The investigators will then study the molecular signaling effect of specific phytocompounds already identified to confer in vivo (mouse), anti-tumor and anti-inflammatory activities, in primary/organoid cultures of human breast tumor cells under ex vivo conditions. Finally, the investigators intend to identify the key molecular regulators, immune-modulatory effectors of test stromal immune cells that are affected by the candidate phytomedicines, using molecular and cell biology assays to investigate the interplay between immune cells and tumor cells in the stromal tissues.

Our study is expected to reveal one or more highly specific, anti-inflammatory phytocompounds that mechanistically confer specific effects on stromal fibroblast or immune cell types, resulting in potent anti-tumor effects on test mammary carcinoma systems. Five Specific Aims are thus designed to investigate the immuno-modulating effects of specific medicinal constituents from TCM materials. The experimental findings obtained from this study would provide insights in the molecular, cellular and signaling mechanisms/effects of several medicinal phytocompounds that may have potential applications in chemoprevention or herbal medicine adjuvant treatment of human breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* adult
* breast cancer patient
* had signed the consent agreement, after your surgery, we will collect the sample from surgically removed breast tissue.

Exclusion Criteria:

* pregnancies
* minor children
* teenagers
* neonates

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 415 (Estimated)
Dates: Start 2010-06; Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ning-Sun Yang, Principal Investigator — Academia Sinica, Taiwan
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan